CLINICAL TRIAL: NCT00038675
Title: Therapy of Hypereosinophilic Syndrome, Polycythemia Vera, Atypical CML or CMML With Platelet Derived Growth Factor (PDGF-R) Fusion Genes, or Mastocytosis With Imatinib Mesylate (STI571)
Brief Title: Therapy of HES, PV, Atypical Chronic Myelocytic Leukemia (CML) or Chronic Myelomonocytic Leukemia (CMML), and Mastocytosis With Imatinib Mesylate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID01-167
Record Dates: First submitted 2002-06-04; First posted 2002-06-05 (Estimated); Results first posted 2022-01-04 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Chronic Myelomonocytic Leukemia; Chronic Myeloid Leukemia; Polycythemia Vera; Hypereosinophilic Syndrome; Mastocytosis
Keywords: Leukemia; Chronic Myelomonocytic Leukemia; Chronic Myeloid Leukemia; Polycythemia Vera; Hypereosinophilic Syndrome; Mastocytosis; Imatinib Mesylate; Gleevec
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Polycythemia Vera; Hypereosinophilic Syndrome; Mastocytosis; Leukemia | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Imatinib (Experimental): Imatinib mesylate 400 mg orally daily, and in HES patients start with imatinib mesylate 100 mg orally daily.
  Interventions: Drug: Imatinib Mesylate (Gleevec)

INTERVENTIONS:
Drug: Imatinib Mesylate (Gleevec) — Imatinib mesylate 400 mg orally daily, and in HES patients start with imatinib mesylate 100 mg orally daily
  Other Names: Gleevec

SUMMARY:
The goal of this clinical research study is to see if Gleevec, known as imatinib mesylate (STI571), can improve the disease condition in patients with hypereosinophilic syndrome, polycythemia vera, atypical CML or CMML with PDGF-R fusion genes, or mastocytosis.

DETAILED DESCRIPTION:
Imatinib mesylate is a chemical compound that blocks a protein that is responsible for a certain form of leukemia. However, imatinib mesylate also blocks other important proteins that may be responsible for other blood diseases such as myeloproliferative disorders.

Patients in this study will take 4 tablets of imatinib mesylate by mouth every day. Patients with HES will take 1 tablet daily to begin, and may go up to 4 tablets daily depending on response. Imatinib mesylate should be taken each morning at breakfast with a large glass of water. Bottles containing the tablets will be given to the patient every month. Unused supplies must be returned at the end of the study. Patients taking oral hydroxyurea to control their blood counts, can continue it during the first month of imatinib mesylate treatment, but must stop taking it from then on.

After completing 2 months of therapy, response to imatinib mesylate will be evaluated. If the response is good, treatment with imatinib mesylate alone will be continued. If the response is not good, the dose of imatinib mesylate will be increased to 8 tablets daily (4 in the morning and 4 in the evening) or may be decreased to 3 tablets daily. This will be based on how the drug is tolerated. Treatment may be continued for up to one year, or as long as it is judged best to control the leukemia.

Patients will be asked to visit their doctor for a physical exam and vital signs. The frequency of doctor visits will vary depending on physical condition.

Blood tests (about 2 teaspoons) will be done once each year. The blood samples will be used for routine lab tests. A bone marrow sample will also be taken to check and measure cells related to the disease after 3 - 4 months, then every 3-6 months in the first year. If the initial bone marrow sample does not show disease, repeated bone marrows will not be done.

This is an investigational study. Imatinib mesylate has been approved in CML for patients whose disease has not responded to interferon. However, this is an investigational study in patients with myeloproliferative diseases. The FDA has authorized the use of imatinib mesylate in research. A total of 145 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have 1 of the following hematopoietic malignancies: Hypereosinophilic syndrome (HES), Polycythemia vera (PV), Atypical CML or CMML with PDGF-R fusion genes, Mastocytosis, Serum bilirubin less than 2 mg%, serum creatinine less than 2 mg% unless abnormality is considered due to hematologic malignancy by investigator, Eastern Cooperative Oncology Group (ECOG) performance status < 3, life expectancy > 12 wks,
2. continued from above. Participants must sign informed consent indicating they are aware of the investigational nature of the study, in keeping with policies of the hospital, women of pregnancy potential must practice birth control. Women and men must continue birth control for the duration of the trial and at least 3 months after the last dose of study drug. Inclusion of women and minorities: As per NIH policy, women and members of minorities will be included as they are referred in the relevant populations.
3. continued from above. There are no exclusions of women or minorities based on the study objectives, New York Heart Association (NYHA) Class <3.

Exclusion Criteria:

N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2001-06; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Cortes, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Official Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All recruitment done at The University of Texas (UT) MD Anderson Cancer Center.
Groups:
- Imatinib Mesylate: Imatinib mesylate 400 mg orally daily, HES participants start with 100 mg orally daily.
Period: Overall Study
Arm/Group | Imatinib Mesylate
Started | 125
Completed | 125
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Imatinib Mesylate
Number analyzed (Participants) | 125
Age, Continuous [Median (Full Range); unit: years] | 56 [21 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 76
Region of Enrollment [Number; unit: participants]
  United States | 125
Leukemia Diagnosis Categories [Number; unit: participants] — Leukemia diagnosis and any subtype determination confirmed via bone marrow aspirate and/or biopsy, assessed prior to treatment.
  participants
    Acute Leukemia | 10
    Chronic myeloproliferative disorders (CMPD) | 7
    Chronic Myelomonocytic Leukemia (CMML) | 11
    Essential Thrombocythemia | 2
    Hypereosinophilic syndrome (HES) | 20
    Systemic mastocytosis (SM) | 25
    Myelodysplastic syndromes (MDS) | 7
    Myelofibrosis | 18
    Polycythemia Vera (PV) | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Complete Response (CR)
Description: Acute myeloid leukemia (AML), Myelodysplastic Syndromes (MDS): CR=Normalization peripheral blood & bone marrow with 5% or less blasts; normo- or hypercellular marrow; Absolute Neutrophil Count (ANC) > 1.0 x 10^9/L, & platelet count >100 x 10^9/L; or CR marrow=As per CR but platelet count < 100 x 10^9/L. Agnogenic myeloid metaplasia (AMM) & CMML: CR=Absence of signs/symptoms of disease; White blood count between 1 to 10 x 10^9/L with no peripheral blasts, promyelocytes, or myelocytes and normalization of bone marrow (< 5% blasts in normocellular or hypercellular marrow) for 4+ weeks. PV: CR=normalization of hemoglobin/hematocrit without need for phlebotomies, disappearance all signs/symptoms of disease. HES: CR=disappearance of eosinophilia (</=10%), disappearance signs/symptoms of disease. Mastocytosis: CR=disappearance of mast cell infiltrates in affected organs, decrease of serum tyrptase levels to <20 ng/ml, & disappearance of SM-associated organomegaly.
Time Frame: after 2 months of therapy, up to 1 year.
Measure: Number; unit: participants
Arm/Group | Imatinib Mesylate
Number analyzed (Participants) | 125
participants
  Acute Leukemia | 0
  Chronic myeloproliferative disorders (CMPD) | 0
  Chronic Myelomonocytic Leukemia (CMML) | 2
  Essential Thrombocythemia | 0
  Hypereosinophilic syndrome (HES) | 3
  Systemic mastocytosis (SM) | 4
  Myelodysplastic syndromes (MDS) | 0
  Myelofibrosis | 1
  Polycythemia Vera (PV) | 2

2. Secondary Outcome: Duration of Response
Description: Time from response to disease progression, measuring length of the response in those participants who responded.
Time Frame: From response evaluation (first evaluation following 2 months therapy) to disease progression or death or until disease progression whichever occurs first, up to 12 years and 5 months
Measure: Median (Full Range); unit: Months
Arm/Group | Imatinib Mesylate
Number analyzed (Participants) | 125
Months | 68 [33.3 to 149]

3. Secondary Outcome: Overall Survival
Description: Overall survival defined as time from registration to disease progression or death from any cause.
Time Frame: From the start of therapy to death or disease progression, assessed up to 12 years and 5 months
Measure: Median (Full Range); unit: Months
Arm/Group | Imatinib Mesylate
Number analyzed (Participants) | 125
Months | 73.2 [0.3 to 149]

ADVERSE EVENTS:
Time Frame: Adverse Event collection from first treatment through 30 days following last treatment, treatment may continue up to one year without disease progression.
Arm/Group | Imatinib Mesylate
All-Cause Mortality (participants affected / at risk) | 10/125
Serious Adverse Events (participants affected / at risk) | 13/125
Other Adverse Events (participants affected / at risk) | 0/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imatinib Mesylate (N=125)
Death (General disorders) | 10 (10)
Hepatic Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Herniated disc Surgery (Surgical and medical procedures) | 1 (1)
GI Hemorrhage (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Second Malignancy (Basal Cell Carcinoma) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes